CLINICAL TRIAL: NCT06628986
Title: the Effect of MBSR and NLP Applications on Fatigue, Sleep Quality, Lactation and Postpartum Depression in the Postpartum Period After Caesarean Section
Brief Title: MBSR and NLP, Postpartum Breastfeeding and Depression
Acronym: postpartum
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aysegul Kilicli (Other)
Responsible Party: Sponsor-Investigator, Aysegul Kilicli, Gaziantep University Health Sciences Institute, Department of Nursing PhD., University of Gaziantep
Organization: University of Gaziantep (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Mauniv
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Breastfeeding, Exclusive; Fatigue; Sleep; Postpartum Depression
Keywords: breastfeeding; fatigue; sleep; postpartum depression
MeSH Terms: conditions — Breast Feeding; Fatigue; Depression, Postpartum | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness-based stress reduction program (Experimental): MBSR; Mindfulness-based stress reduction program. 8 weeks of practice once a week for 20 minutes each. Mindfulness-based stress reduction practices will be carried out online. Mothers will actively participate.
  Interventions: Behavioral: MBSR
- Neurolinguistic programming (Experimental): NLP; Neurolinguistic programming 8 weeks of practice once a week for 20 minutes each. Neurolinguistic programming will be carried out online. Mothers will actively participate.
  Interventions: Behavioral: NLP
- control (Experimental): control; MBSR and NLP applications will not be performed. Mothers will be monitored online every week.
  Interventions: Behavioral: control

INTERVENTIONS:
Behavioral: MBSR — 20 minutes once a week for 8 weeks
  Other Names: MBSR mindfulness-based stress reduction program
  Arms: Mindfulness-based stress reduction program
Behavioral: NLP — NLP Neurolinguistic programming, 20 minutes once a week for 8 weeks
  Other Names: NLP Neurolinguistic programming
  Arms: Neurolinguistic programming
Behavioral: control — control group, no practice,
  Other Names: control group
  Arms: control

SUMMARY:
The postnatal period is a risky period in which mothers experience regressive and progressive changes and rapid biopsychosocial changes. Since this process affects not only the mother but also the family, mothers are under intense stress due to adaptation to the changes that occur in this period.

DETAILED DESCRIPTION:
The postnatal period is a risky period in which retrogressive and progressive changes and rapid biopsychosocial changes occur in mothers. Since this process affects not only the mother but also the family, mothers are under intense stress due to adaptation to the changes occurring in this period. Studies have reported that the most common physical problems in the early postpartum period after caesarean section are pain in the incision area, difficulty in caring for the baby alone, activity intolerance, fatigue, insomnia, breastfeeding problems (such as nipple or lack of milk), mastitis and abdominal tension/gas. As important as it is to reduce postpartum symptoms after caesarean section, it is also important to support and maintain breastfeeding. However, postpartum symptoms such as pain, fatigue and negative effects of anaesthesia after caesarean section negatively affect the breastfeeding process and lead to a delay in the onset of lactation.

When the literature was examined, no study was found that examined the effects of mindfulness-based stress reduction programme and neurolinguistic programme on fatigue, sleep quality, lactation and depression in the postpartum long term.

ELIGIBILITY:
Inclusion Criteria:

* 19-35 years old
* caesarean section
* primiparous
* breastfeeding women

Exclusion Criteria:

* women who refused to participate in the research.

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale for Fatigue (VAS-F) | before the first application
  Visual Analogue Scale for Fatigue (VAS-F), The most positive expression of the fatigue sub-dimension is 0 and the most negative expression is 10, the most negative expression of the energy sub-dimension is 0 and the most positive expression is 10.
Visual Analogue Scale for Fatigue (VAS-F) | Week 4
  Visual Analogue Scale for Fatigue (VAS-F) The most positive expression of the fatigue sub-dimension is 0 and the most negative expression is 10, the most negative expression of the energy sub-dimension is 0 and the most positive expression is 10.
Visual Analogue Scale for Fatigue (VAS-F) | Week 8
  Visual Analogue Scale for Fatigue (VAS-F) The most positive expression of the fatigue sub-dimension is 0 and the most negative expression is 10, the most negative expression of the energy sub-dimension is 0 and the most positive expression is 10.
Pittsburgh Sleep Quality Index (PSQI) | before the first application
  Pittsburgh Sleep Quality Index (PSQI) Each item is evaluated as 0-3 points and the sum of the 7 subcomponents constitutes the PDQI score. The lowest score of the scale is 0 and the highest score is 21. A total PDQI score of ≤5 indicates good sleep and >5 indicates poor sleep.
Pittsburgh Sleep Quality Index (PSQI) | week 4
  Pittsburgh Sleep Quality Index (PSQI) Each item is evaluated as 0-3 points and the sum of the 7 subcomponents constitutes the PDQI score. The lowest score of the scale is 0 and the highest score is 21. A total PDQI score of ≤5 indicates good sleep and >5 indicates poor sleep.
Pittsburgh Sleep Quality Index (PSQI) | week 8
  Pittsburgh Sleep Quality Index (PSQI) Each item is evaluated as 0-3 points and the sum of the 7 subcomponents constitutes the PDQI score. The lowest score of the scale is 0 and the highest score is 21. A total PDQI score of ≤5 indicates good sleep and >5 indicates poor sleep.
Bristol Breastfeeding Assessment Tool (BBAT) | before the first application
  Bristol Breastfeeding Assessment Tool (BBAT) In the scoring of the scale, each item is between 0-2 points. The calculation method is to sum all the scores obtained from the scale items. The lowest score obtained from the scale is 0 and the highest score is 8. The scale does not have a cut-off point. A low score indicates that breastfeeding is not effective and a high score indicates that breastfeeding is effective.
Bristol Breastfeeding Assessment Tool (BBAT) | week 4
  Bristol Breastfeeding Assessment Tool (BBAT) In the scoring of the scale, each item is between 0-2 points. The calculation method is to sum all the scores obtained from the scale items. The lowest score obtained from the scale is 0 and the highest score is 8. The scale does not have a cut-off point. A low score indicates that breastfeeding is not effective and a high score indicates that breastfeeding is effective.
Bristol Breastfeeding Assessment Tool (BBAT) | week 8
  Bristol Breastfeeding Assessment Tool (BBAT) In the scoring of the scale, each item is between 0-2 points. The calculation method is to sum all the scores obtained from the scale items. The lowest score obtained from the scale is 0 and the highest score is 8. The scale does not have a cut-off point. A low score indicates that breastfeeding is not effective and a high score indicates that breastfeeding is effective.
Edinburgh Postpartum Depression Scale (EPDS) | before the first application
  Edinburgh Postpartum Depression Scale (EPDS) The scale is a 4-point Likert-type scale consisting of 10 items. Responses consisting of four options are scored between 0 and 3. A minimum of 0 and a maximum of 30 points can be obtained from the scale. The cut-off point of the scale is 13 points and above for women and 10 points and above for men, and above this point indicates the presence of depression.
Edinburgh Postpartum Depression Scale (EPDS) | week 4
  Edinburgh Postpartum Depression Scale (EPDS) The scale is a 4-point Likert-type scale consisting of 10 items. Responses consisting of four options are scored between 0 and 3. A minimum of 0 and a maximum of 30 points can be obtained from the scale. The cut-off point of the scale is 13 points and above for women and 10 points and above for men, and above this point indicates the presence of depression.
Edinburgh Postpartum Depression Scale (EPDS) | week 8
  Edinburgh Postpartum Depression Scale (EPDS) The scale is a 4-point Likert-type scale consisting of 10 items. Responses consisting of four options are scored between 0 and 3. A minimum of 0 and a maximum of 30 points can be obtained from the scale. The cut-off point of the scale is 13 points and above for women and 10 points and above for men, and above this point indicates the presence of depression.
Breastfeeding Self-Efficacy Scale (BSES) | before the first application
  Breastfeeding Self-Efficacy Scale (BSES) The scale consists of 14 items, five-point Likert type. The items of the scale are evaluated on a scale from '1=never sure' to 5=always sure'. A minimum of 14 points and a maximum of 70 points can be obtained from the scale. All items are positive. The higher the score obtained from the scale, the higher the breastfeeding self-efficacy.
Breastfeeding Self-Efficacy Scale (BSES) | week 4
  Breastfeeding Self-Efficacy Scale (BSES) The scale consists of 14 items, five-point Likert type. The items of the scale are evaluated on a scale from '1=never sure' to 5=always sure'. A minimum of 14 points and a maximum of 70 points can be obtained from the scale. All items are positive. The higher the score obtained from the scale, the higher the breastfeeding self-efficacy.
Breastfeeding Self-Efficacy Scale (BSES) | week 8
  Breastfeeding Self-Efficacy Scale (BSES) The scale consists of 14 items, five-point Likert type. The items of the scale are evaluated on a scale from '1=never sure' to 5=always sure'. A minimum of 14 points and a maximum of 70 points can be obtained from the scale. All items are positive. The higher the score obtained from the scale, the higher the breastfeeding self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: AYŞEGÜL KILIÇLI, Dr., Study Director — Muş Alparslan University
Locations (1):
- Şanlıurfa training and research hospital, Sanliurfa, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 8 October 2024 - 30 October 2025
Access Criteria: 8 October 2024 - 30 October 2025